CLINICAL TRIAL: NCT04432155
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of Xenon Inhalation for Treatment of Patients With Panic Disorder
Brief Title: Xenon Inhalation for Treatment of Panic Disorder
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nobilis Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBTX-002
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Xenon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBTX-001 (Experimental): Combination Product: NBTX-001 Xenon Inhaler The NBTX-001 medical gas consists of 30% xenon, 30% oxygen, and 40% nitrogen. The dose of medical gas is 10 L by volume.
  Interventions: Drug: Xenon
- Placebo (Placebo Comparator): Combination Product: Placebo The placebo medical gas consists of 30% oxygen and 70% nitrogen. The dose of placebo medical gas is 10 L by volume.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xenon — 30% xenon, 30% oxygen, and 40% nitrogen
  Arms: NBTX-001
Drug: Placebo — 30% oxygen, and 70% nitrogen
  Arms: Placebo

SUMMARY:
This study is a double-blind, randomized, placebo-controlled, clinical trial in parallel groups in patients with panic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of panic disorder according to DSM-5.
* Male and female patients ≥18 years of age.

Exclusion Criteria:

* History of schizophrenia, bipolar and other psychotic disorders.
* Patients with underlying pulmonary disease, chronic obstructive pulmonary disease (COPD), asthma, severe lung disease and/or baseline oxygen saturations <92% or any other respiratory conditions / diseases that may affect the respiratory function.
* Currently undergoing targeted empirically-driven psychotherapy for panic disorder or panic disorder-related symptoms.
* Currently undergoing exposure-based psychotherapy for any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
PDSS | Baseline to Week 6
  Panic Disorder Severity Scale

SECONDARY OUTCOMES:
PHQ-9 | Baseline to Week 6
  Patient Health Questionnaire-9

IPD SHARING:
Plan to Share IPD: Undecided